CLINICAL TRIAL: NCT00192699
Title: 10 Year Follow-up Investigation of Patients Who Have Underwent Total Hip Arthroplasty With a Cemented Bi-metric Stem
Brief Title: Bimetric-10: Investigation of Patients Who Have Underwent Total Hip Arthroplasty With a Cemented Bi-Metric Stem
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: ON-04-008b-JPE
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthrosis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: Cemented Bi-Metric femoral stem: Cemented Bi-Metric femoral stem
  Interventions: Device: Bimetric femoral stem

INTERVENTIONS:
Device: Bimetric femoral stem — Cemented Bi-Metric femoral stem
  Other Names: Cemented Bi-Metric femoral stem

SUMMARY:
This is a 10 year follow-up investigation of patients who have underwent total hip arthroplasty with a cemented Bimetric stem.

ELIGIBILITY:
Inclusion criteria:

* Osteoarthrosis

Exclusion criteria:

* Malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarthrosis in hip who have underwent surgery for 10 years ago using Cemented Bi-Metric femoral stem.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2004-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B Laursen, MD, PhD, Principal Investigator — Northern Orthopaedic Division, Aalborg University Hospital, Denmark
Locations (1):
- Northern Orthopaedic Division, Aalborg University Hospital, Aalborg, Northern Jutland, Denmark